CLINICAL TRIAL: NCT02847637
Title: A Randomized, Multicenter, Open-Label, Phase III Clinical Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Prophylactic Emicizumab Versus no Prophylaxis in Hemophilia A Patients Without Inhibitors
Brief Title: A Clinical Trial to Evaluate Prophylactic Emicizumab Versus no Prophylaxis in Hemophilia A Participants Without Inhibitors
Acronym: HAVEN 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH30071; 2016-000072-17 (EudraCT Number)
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Emicizumab
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm C (Control): No Prophylaxis, Then Emicizumab (Active Comparator): Participants who had received episodic treatment with FVIII prior to study entry were randomized to continue episodic FVIII treatment when they started the trial. After completing 24 weeks of no prophylaxis (i.e., episodic FVIII treatment) on study, then they were given the opportunity to switch to emicizumab prophylaxis of 3 mg/kg subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of 3 mg/kg emicizumab SC once every 2 weeks (Q2W). Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
  Interventions: Drug: Emicizumab; Drug: Factor VIII (FVIII)
- Arm A: Emicizumab 1.5 mg/kg QW (Experimental): Participants who had received episodic treatment with FVIII prior to study entry were randomized to receive emicizumab prophylaxis at a dose of 3 milligrams per kilogram (mg/kg) subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of 1.5 mg/kg emicizumab SC QW. Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
  Interventions: Drug: Emicizumab; Drug: Factor VIII (FVIII)
- Arm B: Emicizumab 3 mg/kg Q2W (Experimental): Participants who had received episodic treatment with FVIII prior to study entry were randomized to receive emicizumab prophylaxis at a dose of 3 mg/kg subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of 3 mg/kg emicizumab SC once every 2 weeks (Q2W). Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
  Interventions: Drug: Emicizumab; Drug: Factor VIII (FVIII)
- Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) (Experimental): Participants who had received FVIII prophylaxis prior to study entry were enrolled to receive emicizumab prophylaxis at a dose of 3 mg/kg subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of 1.5 mg/kg emicizumab SC QW. Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
  Interventions: Drug: Emicizumab; Drug: Factor VIII (FVIII)

INTERVENTIONS:
Drug: Emicizumab — Participants received emicizumab prophylaxis subcutaneously at the specified dose for each arm. After at least 24 weeks on prophylactic emicizumab, individuals who experienced suboptimal bleeding control on emicizumab (according to protocol-defined criteria) had the opportunity to increase their dose to 3 mg/kg weekly. Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant had the option to choose a preferred emicizumab dosing regimen among those permitted (i.e., emicizumab 1.5 mg/kg once every week [QW], 3 mg/kg once every 2 weeks [Q2W], or 6 mg/kg once every 4 weeks [Q4W]) and continue on that dosing regimen until discontinuation from the study.
  Other Names: Hemlibra; RO5534262; ACE910
Drug: Factor VIII (FVIII) — FVIII was allowed to treat bleeds on an episodic basis, per the local prescribing information. Specific dosages of FVIII were not mandated in the study. Breakthrough bleeds were to be treated with the lowest FVIII dose expected to achieve hemostasis, which may have been lower than the participant's prior FVIII dose. To avoid bleeds before adequate emicizumab level is reached, patients in Arm D continued their regular FVIII prophylaxis until the second emicizumab loading dose. Concomitant routine FVIII prophylaxis was not permissible otherwise during the study.

SUMMARY:
This is a randomized, global, multicenter, open-label, Phase 3 clinical study in participants with severe hemophilia A without inhibitors against Factor VIII (FVIII) who are 12 years or older. The study evaluates two prophylactic emicizumab regimens versus no prophylaxis in this population with emphasis on efficacy, safety, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >/= 40 kilogram (kg) at the time of screening
* Diagnosis of severe congenital hemophilia A
* Documentation of the details of prophylactic or episodic FVIII treatment and of number of bleeding episodes for at least the last 24 weeks
* Adequate hematologic function
* Adequate hepatic function
* Adequate renal function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 5 elimination half-lives (24 weeks) after the last dose of study drug

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A
* Previous or current treatment for thromboembolic disease or signs of thromboembolic disease
* Conditions that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known human immunodeficiency virus (HIV) infection with cluster of differentiation (CD) 4 count <200 cells per microliter (cells/mcL) within 24 weeks prior to screening. Participants with HIV infection who has CD4 greater than (>) 200 and meet all other criteria are eligible
* Use of systemic immunomodulators at enrollment or planned use during the study, with the exception of anti-retroviral therapy
* Participants who are at high risk for thrombotic microangiopathy (TMA) (for example, have a previous medical or family history of TMA), in the investigator's judgment
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose additional risk, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study
* Planned surgery (excluding minor procedures) during the study
* Receipt of emicizumab in a prior investigational study; an investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration; a non-hemophilia-related investigational drug concurrently, within last 30 days or 5 half-lives, whichever is shorter
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (8):
  - Santa Monica Oncology Center, Santa Monica, California
  - Georgetown Uni Medical Center; Lombardi Cancer Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute; Brigham and Women's Cancer Center, Boston, Massachusetts
  - Children's Hospital of Michigan; Pediatrics, Detroit, Michigan
  - Cornell Univ Medical College; Hematology-Oncolog, New York, New York
  - Bloodworks Northwest (formerly Puget Sound Blood Center); Hemophilia, Seattle, Washington
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne; Thrombosis and Haemostasis Unit, Melbourne, Victoria
  - The Perth Blood Institute, Nedlands, Western Australia
- ICIC, San José, Costa Rica
- France (3):
  - Hopital Cardio-vasculaire Louis Pradel; Hemostase clinique, Bron
  - CH de Bicetre; Centre de Traitement d' Hemophilie, Le Kremlin-Bicêtre
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Universitätsklinikum Bonn; Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn, Germany
- St James's Hospital, Dublin, Ireland
- Italy (2):
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy
  - AOU Careggi; SOD Malattie Emorragiche, Florence, Tuscany
- Japan (7):
  - Nagoya University Hospital, Aichi
  - St. Marianna University Hospital, Kanagawa
  - Sendai Medical Center, Miyagi
  - Nara Medical University Hospital, Nara
  - NHO Osaka National Hospital, Osaka
  - Tokyo Medical University Hospital, Tokyo
  - Ogikubo Hospital, Tokyo
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne; Klinika Hematologii i Transplantologii, Gdansk
  - SPSK Nr1 Klinika Hematoo&Transpl.Szpiku, Lublin
  - ALVAMED Lekarskie Gabinety Specjalistyczne, Poznan
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
- Charlotte Maxeke Johannesburg Hospital; Haemophilia Comprehensive Care Center, Johannesburg, South Africa
- Severance Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
- Taiwan (3):
  - Changhua Christian Hospital, Chang-hua
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
- United Kingdom (2):
  - Cardiff and Vale NHS Trust, Cardiff
  - Royal Free Hospital; Haemophilia Centre, London

REFERENCES:
- [Derived] Kruse-Jarres R, Peyvandi F, Oldenburg J, Chang T, Chebon S, Doral MY, Croteau SE, Lambert T, Kempton CL, Pipe SW, Ko RH, Trzaskoma B, Dhalluin C, Bienz NS, Niggli M, Lehle M, Paz-Priel I, Young G, Jimenez-Yuste V. Surgical outcomes in people with hemophilia A taking emicizumab prophylaxis: experience from the HAVEN 1-4 studies. Blood Adv. 2022 Dec 27;6(24):6140-6150. doi: 10.1182/bloodadvances.2022007458. PMID 35939785
- [Derived] Kiialainen A, Niggli M, Kempton CL, Castaman G, Chang T, Paz-Priel I, Adamkewicz JI, Levy GG. Effect of emicizumab prophylaxis on bone and joint health markers in people with haemophilia A without factor VIII inhibitors in the HAVEN 3 study. Haemophilia. 2022 Nov;28(6):1033-1043. doi: 10.1111/hae.14642. Epub 2022 Jul 29. PMID 35905294
- [Derived] Mahlangu J, Oldenburg J, Paz-Priel I, Negrier C, Niggli M, Mancuso ME, Schmitt C, Jimenez-Yuste V, Kempton C, Dhalluin C, Callaghan MU, Bujan W, Shima M, Adamkewicz JI, Asikanius E, Levy GG, Kruse-Jarres R. Emicizumab Prophylaxis in Patients Who Have Hemophilia A without Inhibitors. N Engl J Med. 2018 Aug 30;379(9):811-822. doi: 10.1056/NEJMoa1803550. PMID 30157389

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 161 participants were screened; 9 failed screening, and 152 participants, who had previously received either episodic or prophylactic treatment with FVIII agents, were enrolled in this study. Participants in Arms C, A, and B were randomized in a 1:2:2 ratio, respectively; participants in Arm D were enrolled without randomization.
Groups:
- Arm C (Control): No Prophylaxis, Then Emicizumab: Participants who had received episodic treatment with FVIII prior to study entry were randomized to continue episodic FVIII treatment when they started the trial. After completing 24 weeks of no prophylaxis (i.e., episodic FVIII treatment) on study, then they were given the opportunity to switch to emicizumab prophylaxis of 3 milligrams per kilogram (mg/kg) subcutaneously (SC) once per week (QW) for 4 weeks followed by maintenance dosing of 3 mg/kg emicizumab SC once every 2 weeks (Q2W). Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
- Arm B: Emicizumab 3 mg/kg Q2W: Participants who had received episodic treatment with FVIII prior to study entry were randomized to receive emicizumab prophylaxis at a dose of 3 milligrams per kilogram (mg/kg) subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of 3 mg/kg emicizumab SC once every 2 weeks (Q2W). Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
Period: Overall Study
Arm/Group | Arm C (Control): No Prophylaxis, Then Emicizumab | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Started | 18 | 36 | 35 | 63
Completed First 24 Weeks of Treatment | 16 (A total of 17 participants in Arm C switched from no prophylaxis to receive emicizumab prophylaxis; however, 1 switched to emicizumab prior to completing 24 weeks on no prophylaxis (at 23.5 weeks).) | 35 | 34 | 63
Emicizumab Dose Was Up-Titrated | 0 | 1 | 1 | 7
Opted to Change Emicizumab Dosing Regimen (Upon Implementation of Protocol Version 4) | 1 | 3 | 1 | 1
Completed | 17 | 34 | 34 | 63
Not Completed | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm C (Control): No Prophylaxis, Then Emicizumab | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | Total
Number analyzed (Participants) | 18 | 36 | 35 | 63 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.9) | 39.8 (14.0) | 40.4 (11.4) | 36.4 (14.4) | 38.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 18 | 36 | 35 | 63 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 5 | 7 | 16
  Not Hispanic or Latino | 17 | 32 | 30 | 53 | 132
  Unknown or Not Reported | 1 | 0 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 6 | 10 | 12 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 3 | 1 | 1 | 8
  White | 11 | 24 | 20 | 47 | 102
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 4 | 3 | 9
Number of Participants with <9 or ≥9 Bleeds in the Last 24 Weeks Prior to Study Entry [Count of Participants; unit: Participants]
  Less Than (<) 9 Bleeds | 4 | 9 | 5 | 53 | 71
  Greater Than or Equal To (≥) 9 Bleeds | 14 | 27 | 30 | 10 | 81
Number of Target Joints in the Last 24 Weeks Prior to Study Entry [Mean (Standard Deviation); unit: target joints] — A target joint was defined as at least 3 bleeds into the same joint over the last 24 weeks prior to study entry.
  target joints | 2.2 (1.4) | 2.1 (1.4) | 2.2 (1.7) | 1.0 (1.6) | 1.7 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR) for Treated Bleeds
Description: The number of treated bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was assessed using a negative binomial (NB) regression model, which accounts for different follow-up times, with the number of bleeds as a function of randomization and the time that each participant stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes the number of bleeds (<9 or ≥9) in the last 24 weeks prior to study entry as a stratification factor. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of the time between treatment and the preceding bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to at least 24 weeks (median [min-max] efficacy periods for Arm C: 24.00 [14.4-25.0] weeks; Arm A: 29.57 [17.3-49.6] weeks; Arm B: 31.29 [3.3-50.6] weeks; Arm D: 33.14 [18.4-48.6] weeks)
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Groups:
- Arm C (Control): No Prophylaxis: Participants who had received episodic treatment with FVIII prior to study entry were randomized to continue episodic FVIII treatment when they started the trial; they were given the opportunity to switch to emicizumab prophylaxis after completing 24 weeks of no prophylaxis. The results for this control arm represent data collected during the first 24 weeks on study while receiving their usual care of episodic treatment with FVIII.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 63
treated bleed rate per year | 38.2 [22.86 to 63.76] | 1.5 [0.89 to 2.47] | 1.3 [0.75 to 2.25] | 1.6 [1.07 to 2.44]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; H0 (null hypothesis): ABR Ratio for Arm A versus Arm C = 1. H1 (alternative hypothesis): ABR Ratio for Arm A versus Arm C ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — Statistical significance is controlled at the 2-sided, 0.05 alpha level. The p-value was obtained via a global model with a 3-level categorical effect for treatment (emicizumab 1.5 mg/kg/week, emicizumab 3 mg/kg/2 weeks, or no prophylaxis); ABR Ratio = 0.04, 95% CI 2-sided [0.020 to 0.075] — Arm A is the numerator and Arm C is the denominator for this ABR Ratio
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; H0 (null hypothesis): ABR Ratio for Arm B versus Arm C = 1. H1 (alternative hypothesis): ABR Ratio for Arm B versus Arm C ≠ 1; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.03, 95% CI 2-sided [0.017 to 0.066] — Arm B is the numerator and Arm C is the denominator for this ABR Ratio

2. Secondary Outcome: Annualized Bleeding Rate (ABR) for All Bleeds
Description: The number of all bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was assessed using a NB regression model, which accounts for different follow-up times, with the patient's number of bleeds as a function of randomization and the time that each patient stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes the number of bleeds (<9 or ≥9) in the last 24 weeks prior to study entry as a stratification factor. "All bleeds" comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 63
all bleed rate per year | 47.6 [28.45 to 79.59] | 2.5 [1.63 to 3.90] | 2.6 [1.63 to 4.29] | 3.3 [2.22 to 4.83]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.05, 95% CI 2-sided [0.028 to 0.099] — Arm A is the numerator and Arm C is the denominator for this ABR Ratio
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 1, analysis 1]; ABR Ratio = 0.06, 95% CI 2-sided [0.030 to 0.103] — Arm B is the numerator and Arm C is the denominator for this ABR Ratio

3. Secondary Outcome: Annualized Bleeding Rate (ABR) for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was assessed using a NB regression model, which accounts for different follow-up times, with the patient's number of bleeds as a function of randomization and the time that each patient stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes the number of bleeds (<9 or ≥9) in the last 24 weeks prior to study entry as a stratification factor. A "joint bleed" is defined as a bleed reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint; and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. It is considered a "treated joint bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed". Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 63
treated joint bleed rate per year | 26.5 [14.67 to 47.79] | 1.1 [0.59 to 1.89] | 0.9 [0.44 to 1.67] | 1.2 [0.70 to 2.01]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Stratified Wald test — Statistical significance is controlled at the 2-sided, 0.05 alpha level. The p-value is obtained via a global model with a 3-level categorical effect for treatment (emicizumab 1.5 mg/kg/week, emicizumab 3 mg/kg/2 weeks, or no prophylaxis); ABR Ratio = 0.04, 95% CI 2-sided [0.019 to 0.085] — Arm A is the numerator and Arm C is the denominator for this ABR Ratio
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 3, analysis 1]; ABR Ratio = 0.03, 95% CI 2-sided [0.015 to 0.070] — Arm B is the numerator and Arm C is the denominator for this ABR Ratio

4. Secondary Outcome: Annualized Bleeding Rate (ABR) for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was assessed using a NB regression model, which accounts for different follow-up times, with the patient's number of bleeds as a function of randomization and the time that each patient stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes the number of bleeds (<9 or ≥9) in the last 24 weeks prior to study entry as a stratification factor. A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed". Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 63
treated spontaneous bleed rate per year | 15.6 [7.60 to 31.91] | 1.0 [0.48 to 1.91] | 0.3 [0.11 to 0.75] | 0.5 [0.23 to 0.94]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 3, analysis 1]; ABR Ratio = 0.06, 95% CI 2-sided [0.025 to 0.151] — Arm A is the numerator and Arm C is the denominator for this ABR Ratio
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Stratified Wald test — [p-value comment as in outcome 3, analysis 1]; ABR Ratio = 0.02, 95% CI 2-sided [0.006 to 0.056] — Arm B is the numerator and Arm C is the denominator for this ABR Ratio

5. Secondary Outcome: Annualized Bleeding Rate (ABR) for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period is presented as an annualized bleeding rate (ABR) that was assessed using a NB regression model, which accounts for different follow-up times, with the patient's number of bleeds as a function of randomization and the time that each patient stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes the number of bleeds (<9 or ≥9) in the last 24 weeks prior to study entry as a stratification factor. A "target joint bleed" is defined as a bleed reported as a joint bleed into a target joint, defined as at least 3 bleeds into the same joint during the last 24 weeks prior to study entry. It is considered a "treated target joint bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed". Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: All participants, which includes those randomized to Arms A, B, and C, and those enrolled in Arm D of the study.
Measure: Number (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 63
treated target joint bleed rate per year | 13.0 [5.22 to 32.33] | 0.6 [0.28 to 1.42] | 0.7 [0.27 to 1.64] | 0.6 [0.26 to 1.53]
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Stratified Wald test — Not controlled for type I error; ABR Ratio = 0.05, 95% CI 2-sided [0.016 to 0.143] — Arm A is the numerator and Arm C is the denominator for this ABR Ratio
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Stratified Wald test — Not controlled for type I error; ABR Ratio = 0.05, 95% CI 2-sided [0.018 to 0.147] — Arm B is the numerator and Arm C is the denominator for this ABR Ratio

6. Secondary Outcome: Intra-Participant Comparison of ABR for Treated Bleeds on Study Versus Pre-Study in Participants From the Non-Interventional Study Population Previously Treated With Factor VIII (FVIII) Prophylaxis (NISP)
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for treated bleeds on study versus pre-study in the NIS population previously treated with FVIII prophylaxis in NIS BH29768. The number of treated bleeds over the efficacy period is presented as an ABR that was assessed using a NB regression model, which accounts for different follow-up times, with the number of bleeds as a function of treatment and the time that each participant stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes a repeated statement to account for intra-participant comparison. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of the time between treatment and the preceding bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: Efficacy periods: At least 24 weeks prior to study entry (median [min-max] for Dnisp-FVIII Prophylaxis: 30.07 [5.0-45.1] weeks); and From Baseline to at least 24 weeks on study (median [min-max] for Dnisp-Emicizumab Prophylaxis: 33.71 [20.1-48.6] weeks)
Population: Intra-participant comparison in the NIS population previously treated with FVIII prophylaxis (NISP), which includes all participants who had received FVIII prophylaxis in NIS BH29768 prior to study entry in Arm D.
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Groups:
- Dnisp: Pre-Study FVIII Prophylaxis in NIS BH29768: This arm includes historical data from participants in the non-interventional study (NIS) BH29768 who had received FVIII prophylaxis and were followed for a minimum of 24 weeks on the NIS prior to enrollment in Arm D of this study.
- Dnisp: Emicizumab Prophylaxis (Pre-Study FVIII Prophylaxis): This arm includes data from the same participants who had received FVIII prophylaxis in NIS BH29768 prior to study entry and then enrolled in Arm D of this study to receive emicizumab prophylaxis at a dose of 3 mg/kg once per week (QW) subcutaneously (SC) for 4 weeks, followed by maintenance dosing of 1.5 mg/kg emicizumab SC QW until the end of study. The data reported was collected only during emicizumab prophylaxis treatment.
Arm/Group | Dnisp: Pre-Study FVIII Prophylaxis in NIS BH29768 | Dnisp: Emicizumab Prophylaxis (Pre-Study FVIII Prophylaxis)
Number analyzed (Participants) | 48 | 48
treated bleed rate per year | 4.8 [3.22 to 7.09] | 1.5 [0.98 to 2.33]
Statistical Analysis 1: Comparison: Dnisp: Pre-Study FVIII Prophylaxis in NIS BH29768 vs Dnisp: Emicizumab Prophylaxis (Pre-Study FVIII Prophylaxis); H0 (null hypothesis): ABR Ratio = 1. H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Non-stratified Wald test — Statistical significance is controlled at the 2-sided, 0.05 alpha level; ABR Ratio = 0.32, 95% CI 2-sided [0.195 to 0.514] — Dnisp: Emicizumab Prophylaxis is the numerator and Dnisp: Pre-Study FVIII Prophylaxis is the denominator for this ABR ratio

7. Secondary Outcome: Intra-Participant Comparison of ABR for All Bleeds on Study Versus Pre-Study in Participants From the Non-Interventional Study Population Previously Treated With FVIII Prophylaxis (NISP)
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for all bleeds on study versus pre-study in the NIS population previously treated with FVIII prophylaxis in NIS BH29768. The number of all bleeds over the efficacy period is presented as an ABR that was assessed using a NB regression model, which accounts for different follow-up times, with the participant's number of bleeds as a function of treatment and the time that each participant stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes a repeated statement to account for intra-participant comparison. "All bleeds" comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Dnisp: Pre-Study FVIII Prophylaxis in NIS BH29768 | Dnisp: Emicizumab Prophylaxis (Pre-Study FVIII Prophylaxis)
Number analyzed (Participants) | 48 | 48
all bleed rate per year | 8.9 [5.72 to 13.87] | 3.3 [2.17 to 5.06]
Statistical Analysis 1: Comparison: Dnisp: Pre-Study FVIII Prophylaxis in NIS BH29768 vs Dnisp: Emicizumab Prophylaxis (Pre-Study FVIII Prophylaxis); H0 (null hypothesis): ABR Ratio = 1. H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p = 0.0002, Non-stratified Wald test — Statistical significance is controlled at the 2-sided, 0.05 alpha level; ABR Ratio = 0.37, 95% CI 2-sided [0.220 to 0.626] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Intra-Participant Comparison of ABR for Treated Bleeds on Study Versus Pre-Study in Participants From the NIS Population Previously Treated With Episodic FVIII (NISE)
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for treated bleeds on study versus pre-study in the NIS population previously treated with episodic FVIII in NIS BH29768. The number of treated bleeds over the efficacy period is presented as an ABR that was assessed using a NB regression model, which accounts for different follow-up times, with the number of bleeds as a function of treatment and the time that each participant stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes a repeated statement to account for intra-participant comparison. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of the time between treatment and the preceding bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: Efficacy periods: At least 24 weeks prior to study entry (median [min-max] for A+Bnise-FVIII Episodic: 25.71 [15.4-40.9] weeks); and From Baseline to at least 24 weeks on study (median [min-max] for A+Bnise-Emicizumab: 34.71 [24.1-50.6] weeks)
Population: Intra-participant comparison in the NIS population previously treated with episodic FVIII (NISE), which includes all participants who had received episodic FVIII in NIS BH29768 prior to study entry in Arms A and B (pooled data).
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Groups:
- A+Bnise: Pre-Study Episodic FVIII in NIS BH29768: This arm includes historical data from participants in the non-interventional study (NIS) BH29768 who had received episodic FVIII treatment and were followed for a minimum of 24 weeks on the NIS prior to randomization to Arms A or B of this study. A pooled analysis, as opposed to two separate analyses, was performed due to the small number of NIS episodic patients (NISE) randomized to either Arm A or B.
- A+Bnise: Emicizumab Prophylaxis (Pre-study Episodic FVIII): This arm includes data from the same participants who had received episodic FVIII treatment in NIS BH29768 prior to study entry and then were randomized to Arms A or B of this study to receive emicizumab prophylaxis at a dose of 3 mg/kg subcutaneously (SC) once per week (QW) for 4 weeks, followed by maintenance dosing of either 1.5 mg/kg emicizumab SC QW (Arm A) or 3 mg/kg emicizumab SC Q2W (Arm B). A pooled analysis, as opposed to two separate analyses, was performed due to the small number of NIS episodic patients (NISE) randomized to either Arm A or B. The data reported was collected only during emicizumab prophylaxis treatment.
Arm/Group | A+Bnise: Pre-Study Episodic FVIII in NIS BH29768 | A+Bnise: Emicizumab Prophylaxis (Pre-study Episodic FVIII)
Number analyzed (Participants) | 20 | 20
treated bleed rate per year | 34.4 [27.45 to 43.14] | 1.0 [0.43 to 2.54]
Statistical Analysis 1: Comparison: A+Bnise: Pre-Study Episodic FVIII in NIS BH29768 vs A+Bnise: Emicizumab Prophylaxis (Pre-study Episodic FVIII); H0 (null hypothesis): ABR Ratio = 1. H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Non-stratified Wald test — Not controlled for type I error; ABR Ratio = 0.03, 95% CI 2-sided [0.014 to 0.067] — Arm A+Bnise: Emicizumab Prophylaxis is the numerator and Arm A+Bnise: Pre-Study Episodic FVIII is the denominator for this ABR Ratio

9. Secondary Outcome: Intra-Participant Comparison of ABR for All Bleeds on Study Versus Pre-Study in Participants From the NIS Population Previously Treated With Episodic FVIII (NISE)
Description: This is an intra-participant comparison of the annualized bleeding rate (ABR) for all bleeds on study versus pre-study in the NIS population previously treated with episodic FVIII in NIS BH29768. The number of all bleeds over the efficacy period is presented as an ABR that was assessed using a NB regression model, which accounts for different follow-up times, with the participant's number of bleeds as a function of treatment and the time that each participant stays in the study (i.e., length of the efficacy period) included as an offset in the model. The model also includes a repeated statement to account for intra-participant comparison. "All bleeds" comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | A+Bnise: Pre-Study Episodic FVIII in NIS BH29768 | A+Bnise: Emicizumab Prophylaxis (Pre-study Episodic FVIII)
Number analyzed (Participants) | 20 | 20
all bleed rate per year | 39.6 [31.94 to 49.04] | 1.6 [0.85 to 2.92]
Statistical Analysis 1: Comparison: A+Bnise: Pre-Study Episodic FVIII in NIS BH29768 vs A+Bnise: Emicizumab Prophylaxis (Pre-study Episodic FVIII); H0 (null hypothesis): ABR Ratio = 1. H1 (alternative hypothesis): ABR Ratio ≠ 1; Test type: Superiority; p < 0.0001, Non-stratified Wald test — Not controlled for type I error; ABR Ratio = 0.04, 95% CI 2-sided [0.023 to 0.068] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Hemophilia A Quality of Life (Haem-A-QoL) Questionnaire Physical Health Subscore for Adult Participants (≥18 Years of Age) in the Randomized Population at Week 25
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Physical Health domain score is reported (range 0 to 100, with lower scores reflective of better physical health). The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline, Week 25
Population: Adult participants randomized to Arms A, B, and C. The number analyzed represents participants who provided responses at Baseline and Week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 13 | 34 | 29
units on a scale | 44.32 (17.15) | 31.81 (27.86) | 28.35 (25.57)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; Test type: Superiority; p = 0.0891, ANCOVA — Statistical significance is controlled at the 2-sided, 0.05 alpha level; Mean Difference (Final Values) = 12.51, 95% CI 2-sided [-1.96 to 26.98] — The difference in adjusted means was analyzed as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; Test type: Superiority; p = 0.0349, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = 15.97, 95% CI 2-sided [1.16 to 30.78] — The difference in adjusted means was analyzed as Arm C minus Arm B

11. Secondary Outcome: Haem-A-QoL Questionnaire Total Score for Adult Participants (≥18 Years of Age) in the Randomized Population at Week 25
Description: The Haem-A-QoL questionnaire has been developed and used in hemophilia A participants, assessing very specific aspects of dealing with hemophilia. The questionnaire consists of items pertaining to 10 domains: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain ranges from 0 to 100 with lower scores reflective of better quality of life. Haem-A-QoL Total Score is the average of all domain scores and it ranges from 0 to 100, with lower scores reflective of better quality of life. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline, Week 25
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 13 | 34 | 29
units on a scale | 29.95 (13.56) | 24.04 (15.26) | 21.39 (12.64)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; Test type: Superiority; p = 0.1269, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = 5.91, 95% CI 2-sided [-1.72 to 13.55] — The difference in adjusted means was analyzed as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; Test type: Superiority; p = 0.0317, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = 8.56, 95% CI 2-sided [0.77 to 16.35] — The difference in adjusted means was analyzed as Arm C minus Arm B

12. Secondary Outcome: European Quality of Life 5-Dimensions-5 Levels (EQ-5D-5L) Questionnaire Visual Analogue Scale (VAS) Score in the Randomized Population at Week 25
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline, Week 25
Population: Participants randomized to Arms A, B, and C. The number analyzed represents participants who provided responses at Baseline and Week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 14 | 34 | 29
units on a scale | 72.57 (8.20) | 76.61 (20.99) | 81.72 (15.55)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; Test type: Superiority; p = 0.3402, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = -4.04, 95% CI 2-sided [-12.43 to 4.35] — The difference in adjusted means was analyzed as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; Test type: Superiority; p = 0.0373, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = -9.15, 95% CI 2-sided [-17.74 to -0.55] — The difference in adjusted means was analyzed as Arm C minus Arm B

13. Secondary Outcome: EQ-5D-5L Questionnaire Index Utility Score in the Randomized Population at Week 25
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L VAS. The EQ-5D-5L health state profile is designed to record the participant's current health state in 5 domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. Responses from the five domains are used to calculate a single index utility score on a scale of 0 to 1, with higher scores reflective of better quality of life. The means were derived via an analysis of covariance (ANCOVA) model and have been adjusted for the following co-variates: baseline score, treatment group, and treatment by baseline interaction term.
Time Frame: Baseline, Week 25
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 14 | 34 | 29
units on a scale | 0.63 (0.20) | 0.76 (0.24) | 0.76 (0.18)
Statistical Analysis 1: Comparison: Arm C (Control): No Prophylaxis vs Arm A: Emicizumab 1.5 mg/kg QW; Test type: Superiority; p = 0.0060, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.22 to -0.04] — The difference in adjusted means was analyzed as Arm C minus Arm A
Statistical Analysis 2: Comparison: Arm C (Control): No Prophylaxis vs Arm B: Emicizumab 3 mg/kg Q2W; Test type: Superiority; p = 0.0059, ANCOVA — Not controlled for type I error; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.23 to -0.04] — The difference in adjusted means was analyzed as Arm C minus Arm B

14. Secondary Outcome: Hemophilia-Specific Quality of Life - Short Form (Haemo-QoL-SF) Questionnaire Score in Adolescent Participants (12 to 17 Years of Age) in the Randomized Population at Week 25
Description: The Haemo-QoL-SF contains 35 items, which cover nine domains considered relevant for the children's health-related quality of life (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia and treatment). Items are rated with five respective response options: never, seldom, sometimes, often, and always. Haemo-QoL-SF total score range from 0 to 100, where lower scores reflect better health-related quality of life.
Time Frame: Week 25
Population: The pre-specified efficacy objective was the comparison of Haemo-QoL-SF scores at Week 25 in adolescents who were previously on episodic treatment (i.e., randomized to Arms A, B, or C). Because there was a total of just one adolescent randomized to this study (in Arm C), statistical analyses could not be performed and no data is reported.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants With at Least One Adverse Event During the First 24 Weeks of the Study, Primary Analysis
Description: The percentage of participants experiencing at least one adverse event, including all non-serious and serious adverse events, is reported here. At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: From Baseline to at least 24 weeks (median [min-max] safety periods for Arm C (Control): 24.00 [14.4-25.0] weeks; Arm A: 30.00 [21.4-49.6] weeks; Arm B: 31.29 [24.4-50.6] weeks; Arm C (Emi): 7.57 [0.3-26.3] weeks; Arm D: 33.71 [18.4-49.6] weeks)
Population: All participants in Arms A, B, and D who received at least one dose of emicizumab and all participants in Arm C (Control) who started the no prophylaxis study period. Participants in Arm C (Emi) are those from Arm C who switched after 24 weeks no prophylaxis to receive emicizumab prophylaxis (2 were excluded who did not switch at the time of analysis).
Measure: Number; unit: percentage of participants
Groups:
- Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD): This arm includes all participants from Arm C who had switched to emicizumab prophylaxis up to the primary completion date (PCD; i.e., analysis cutoff) after having completed 24 weeks on No Prophylaxis. The data reported was collected only during emicizumab prophylaxis treatment up to the PCD. Emicizumab was administered at a loading dose of 3 mg/kg SC once per week (QW) for the first 4 weeks, followed by maintenance dosing of 3 mg/kg emcizumab SC Q2W.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 33.3 | 94.4 | 85.7 | 50.0 | 87.3

16. Secondary Outcome: Percentage of Participants With at Least One Grade ≥3 Adverse Event During the First 24 Weeks of the Study, Primary Analysis
Description: The World Health Organization (WHO) toxicity grading scale will be used for assessing adverse event severity. For adverse events that are not specifically listed in the WHO toxicity grading scale, a grade 3 adverse event is defined as: severe, marked limitation in activity, some assistance usually required, medical intervention or therapy required, hospitalization possible; and a grade 4 adverse event is defined as: life-threatening, extreme limitation in activity, significant assistance required, significant medical intervention or therapy required, hospitalization or hospice care probable. At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 5.6 | 8.3 | 11.4 | 0 | 9.3

17. Secondary Outcome: Percentage of Participants With at Least One Adverse Event Leading to Withdrawal From Treatment During the First 24 Weeks of the Study, Primary Analysis
Description: At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 2.9 | 0 | 0

18. Secondary Outcome: Percentage of Participants With at Least One Adverse Event of Changes From Baseline in Vital Signs During the First 24 Weeks of the Study, Primary Analysis
Description: The percentage of participants with adverse events of changes from baseline in vital signs is reported here. Vital signs measurements consisted of heart and respiratory rate, temperature, and systolic and diastolic blood pressures, with an abnormal vital sign value being outside of the normal range. An abnormal vital sign result is reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment (e.g., dosage modification, treatment interruption or discontinuation); results in a medical intervention or a change in concomitant therapy; or is clinically significant in the investigator's judgment. At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With at Least One Adverse Event of Changes From Baseline in Physical Examination Findings During the First 24 Weeks of the Study, Primary Analysis
Description: Post-baseline physical examination abnormalities that were not present at baseline or worsened were reported as adverse events. At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With at Least One Adverse Event of Abnormal Laboratory Values During the First 24 Weeks of the Study, Primary Analysis
Description: The percentage of participants with adverse events of abnormal laboratory values is reported here. An abnormal laboratory value is defined as a laboratory test result outside of the normal range for hematology or serum chemistries. It is reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment (e.g., dosage modification, treatment interruption or discontinuation); results in a medical intervention or a change in concomitant therapy; or is clinically significant in the investigator's judgment. At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 5.6 | 17.1 | 6.3 | 4.8

21. Secondary Outcome: Percentage of Participants With at Least One Local Injection-Site Reaction During the First 24 Weeks of the Study, Primary Analysis
Description: Local adverse events that occurred within 24 hours after study drug administration and, in the investigator's opinion, were judged to be related to study drug injection, were captured as an "injection-site reaction" on the Adverse Event electronic Case Report Form (eCRF). An injection-related reaction that was localized was marked as a "local injection-site reaction." At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 25.0 | 20.0 | 12.5 | 33.3

22. Secondary Outcome: Percentage of Participants With at Least One Thromboembolic Event During the First 24 Weeks of the Study, Primary Analysis
Description: At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of approximately 1 year.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Percentage of Participants With at Least One Thrombotic Microangiopathy During the First 24 Weeks of the Study, Primary Analysis
Description: At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Percentage of Participants With at Least One Systemic Hypersensitivity, Anaphylaxis, or Anaphylactoid Reaction During the First 24 Weeks of the Study, Primary Analysis
Description: At the clinical cut-off date for primary analysis (15 Sep 2017), data was collected over a period of at least 24 weeks.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis up to PCD) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
Number analyzed (Participants) | 18 | 36 | 35 | 16 | 63
percentage of participants | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Safety Summary of the Percentage of Emicizumab-Treated Participants With at Least One Adverse Event During the Study
Description: Investigators sought information on adverse events (AEs) at each contact with participants. The WHO toxicity grading scale was used for assessing AE severity (i.e., intensity of an AE); any AEs not specifically listed in the WHO toxicity grading scale were assessed for severity according to the following grades: Grade 1 is mild; Grade 2 is moderate, Grade 3 is severe; Grade 4 is life-threatening; and Grade 5 is death. Regardless of severity, some AEs may have also met seriousness criteria. The terms "severe" and "serious" are not synonymous; severity and seriousness were independently assessed for each AE. For participants whose emicizumab dose was up-titrated and those who opted for a change in dosing regimen (after implementation of protocol v4), only AEs that occurred before either one of those events are included. Hypersens.= hypersensitivity; Mod. = modification
Time Frame: From start of emicizumab treatment to study completion, dose up-titration, or change of dosing regimen (median [min-max] efficacy period for all emicizumab participants: 228.14 [7.3-288.3] weeks)
Population: All Emicizumab Participants, which includes all participants who received emicizumab on the study. For Arm C (Emi), it only includes participants who crossed over to receive prophylactic treatment with emicizumab after first completing 24 weeks of no prophylaxis on study (1 participant was excluded because they were lost to follow-up before Week 24 and did not receive emicizumab).
Measure: Number; unit: percentage of participants
Groups:
- Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis): This arm includes all participants from Arm C who switched to emicizumab prophylaxis after completing 24 weeks on No Prophylaxis. The data reported was collected only during emicizumab prophylaxis treatment. Emicizumab was administered at a loading dose of 3 mg/kg/week SC for the first 4 weeks (after at least 24 weeks) followed by a maintenance dose of 3 mg/kg once every 2 weeks SC. Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
- All Emicizumab Participants: This analysis set included all participants who received emicizumab on the study. For Arm C, it only includes all participants starting after Week 24 on study when they crossed over to first receive prophylactic treatment with emicizumab.
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
percentage of participants
  Any Adverse Event (AE) | 100.0 | 97.1 | 88.2 | 100.0 | 98.0
  AE with Fatal Outcome | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Serious AE | 27.8 | 22.9 | 5.9 | 25.4 | 23.2
  AE Leading to Withdrawal from Treatment | 0.0 | 2.9 | 0.0 | 0.0 | 0.7
  AE Leading to Dose Mod./Interruption | 2.8 | 0.0 | 0.0 | 1.6 | 1.3
  Grade ≥3 AE | 36.1 | 28.6 | 5.9 | 20.6 | 24.5
  Related AE | 30.6 | 34.3 | 23.5 | 47.6 | 37.7
  Local Injection Site Reaction | 27.8 | 22.9 | 23.5 | 39.7 | 31.1
  Systemic Hypersens./Anaphylac(tic/toid) Reaction | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Thromboembolic Event (TE) | 0.0 | 2.9 | 0.0 | 1.6 | 1.3
  Thrombotic Microangiopathy (TMA) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

26. Secondary Outcome: Long-Term Efficacy of Emicizumab: Model-Based Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Emicizumab Participants
Description: The number of bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (≥) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration or change of dosing regimen were excluded.
Time Frame: as for outcome 25
Population: All Emicizumab Participants, which includes all participants who received emicizumab on the study. For Arm C, it only includes participants who crossed over to receive prophylactic treatment with emicizumab after first completing 24 weeks of no prophylaxis on study.
Measure: Number (95% Confidence Interval); unit: bleeds per year
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
bleeds per year
  Treated Bleeds | 0.8 [0.48 to 1.29] | 0.7 [0.40 to 1.08] | 1.2 [0.47 to 3.19] | 1.5 [1.02 to 2.34] | 1.2 [0.92 to 1.56]
  All Bleeds | 1.1 [0.72 to 1.66] | 1.1 [0.73 to 1.73] | 2.2 [1.16 to 4.15] | 2.4 [1.68 to 3.43] | 1.8 [1.46 to 2.29]
  Treated Spontaneous Bleeds | 0.5 [0.23 to 1.03] | 0.2 [0.10 to 0.45] | 0.4 [0.12 to 1.35] | 0.5 [0.30 to 0.78] | 0.4 [0.29 to 0.58]
  Treated Joint Bleeds | 0.4 [0.24 to 0.73] | 0.4 [0.21 to 0.68] | 0.7 [0.25 to 1.66] | 1.0 [0.60 to 1.76] | 0.7 [0.53 to 1.00]
  Treated Target Joint Bleeds | 0.2 [0.11 to 0.43] | 0.2 [0.08 to 0.39] | 0.4 [0.13 to 1.31] | 0.6 [0.26 to 1.42] | 0.4 [0.29 to 0.66]

27. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Emicizumab Participants
Description: The number of bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (≥) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration or change of dosing regimen were excluded.
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Mean (95% Confidence Interval); unit: bleeds per year
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
bleeds per year
  Treated Bleeds | 1.2 [0.04 to 5.83] | 0.8 [0.01 to 5.23] | 1.2 [0.05 to 5.95] | 1.7 [0.15 to 6.69] | 1.3 [0.07 to 6.07]
  All Bleeds | 1.4 [0.09 to 6.29] | 1.3 [0.07 to 6.10] | 2.2 [0.32 to 7.58] | 2.6 [0.45 to 8.15] | 2.0 [0.23 to 7.19]
  Treated Spontaneous Bleeds | 0.7 [0.00 to 4.97] | 0.3 [0.00 to 4.22] | 0.4 [0.00 to 4.48] | 0.6 [0.00 to 4.81] | 0.5 [0.00 to 4.68]
  Treated Joint Bleeds | 0.6 [0.00 to 4.94] | 0.5 [0.00 to 4.64] | 0.6 [0.00 to 4.95] | 1.1 [0.04 to 5.78] | 0.8 [0.01 to 5.23]
  Treated Target Joint Bleeds | 0.4 [0.00 to 4.54] | 0.3 [0.00 to 4.28] | 0.4 [0.00 to 4.50] | 0.6 [0.00 to 4.92] | 0.5 [0.00 to 4.64]

28. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Emicizumab Participants
Description: as for outcome 27
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: bleeds per year
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
bleeds per year
  Treated Bleeds | 0.4 [0.00 to 1.28] | 0.4 [0.00 to 1.06] | 0.0 [0.00 to 2.48] | 0.5 [0.00 to 1.07] | 0.4 [0.00 to 1.15]
  All Bleeds | 0.5 [0.09 to 1.77] | 0.8 [0.23 to 1.92] | 1.6 [0.20 to 3.8] | 1.0 [0.38 to 2.70] | 1.0 [0.19 to 2.37]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 0.51] | 0.0 [0.00 to 0.23] | 0.0 [0.00 to 0.65] | 0.0 [0.00 to 0.48] | 0.0 [0.00 to 0.40]
  Treated Joint Bleeds | 0.2 [0.00 to 0.89] | 0.2 [0.00 to 0.49] | 0.0 [0.00 to 1.09] | 0.0 [0.00 to 0.59] | 0.2 [0.00 to 0.72]
  Treated Target Joint Bleeds | 0.1 [0.00 to 0.55] | 0.0 [0.00 to 0.37] | 0.0 [0.00 to 0.81] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.38]

29. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: The number of treated bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v4), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: 1-12, 13-24, 25-36, 37-48, 49-60, 61-72, 73-84, 85-96, 97-108, 109-120, 121-132, 133-144, 145-156, 157-168, 169-180, 181-192, 193-204, 205-216, 217-228, 229-240, 241-252, 253-264, 265-276, and 277-288 weeks
Population: All Emicizumab Participants, which includes all participants who received emicizumab on the study. The number analyzed includes participants with available data over each interval.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
Treated bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 1.9 [0.21 to 7.04]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 1.9 [0.20 to 6.99]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 1.0 [0.02 to 5.57]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 0.9 [0.01 to 5.35]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 1.0 [0.02 to 5.54]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 1.1 [0.04 to 5.72]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 0.7 [0.01 to 5.12]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 1.1 [0.03 to 5.68]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 0.9 [0.01 to 5.32]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.6 [0.00 to 4.83]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.5 [0.00 to 4.72]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 1.1 [0.03 to 5.68]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 1.1 [0.03 to 5.70]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 1.1 [0.04 to 5.78]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 1.3 [0.06 to 6.05]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 1.0 [0.02 to 5.56]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 1.6 [0.13 to 6.57]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 0.8 [0.01 to 5.15]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.5 [0.00 to 4.59]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.8 [0.01 to 5.30]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.3 [0.00 to 4.21]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.5 [0.00 to 4.72]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.2 [0.00 to 4.09]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

30. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: Treated bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
Treated bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 0.0 [0.00 to 4.35]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 0.0 [0.00 to 2.17]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.0 [0.00 to 0.00]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.0 [0.00 to 0.00]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.0 [0.00 to 0.00]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [0.00 to 0.00]

31. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: The number of all bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v4), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: All bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
All bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 3.8 [0.97 to 9.91]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 2.8 [0.53 to 8.45]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 1.8 [0.17 to 6.83]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 1.4 [0.10 to 6.33]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 1.5 [0.10 to 6.37]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 1.6 [0.14 to 6.66]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 1.2 [0.05 to 5.88]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 1.4 [0.09 to 6.30]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 1.3 [0.06 to 6.02]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.8 [0.01 to 5.21]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.8 [0.01 to 5.20]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 1.2 [0.04 to 5.84]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 1.3 [0.06 to 6.02]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 1.4 [0.09 to 6.28]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 1.7 [0.15 to 6.72]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 1.4 [0.08 to 6.19]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 1.7 [0.16 to 6.74]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 1.1 [0.04 to 5.72]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.6 [0.00 to 4.91]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.9 [0.02 to 5.41]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.4 [0.00 to 4.47]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.6 [0.00 to 4.86]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.2 [0.00 to 4.09]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

32. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: as for outcome 31
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: All bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
All bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 0.0 [0.00 to 4.35]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 0.0 [0.00 to 4.35]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 0.0 [0.00 to 4.35]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.0 [0.00 to 0.00]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.0 [0.00 to 0.00]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.0 [0.00 to 0.00]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [0.00 to 0.00]

33. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleeding Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: The number of treated spontaneous bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated spontaneous bleeds were defined as treated (with coagulation factors) bleeds with no known contributing factor (e.g., trauma, surgery). The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants with dose up-titration or a change in emicizumab dosing regimen (after implementation of protocol v4), the efficacy period ended the day before the first day on the up-titrated dose or changed dosing regimen.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Mean (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
Treated spontaneous bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 0.7 [0.00 to 4.98]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 0.7 [0.00 to 5.00]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 0.3 [0.00 to 4.30]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 0.4 [0.00 to 4.53]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 0.5 [0.00 to 4.60]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 0.3 [0.00 to 4.25]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 0.1 [0.00 to 3.95]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 0.4 [0.00 to 4.48]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 0.2 [0.00 to 4.14]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.2 [0.00 to 4.03]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.1 [0.00 to 3.96]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 0.6 [0.00 to 4.78]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 0.6 [0.00 to 4.87]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 0.2 [0.00 to 4.09]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 0.4 [0.00 to 4.50]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 0.2 [0.00 to 4.01]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 0.1 [0.00 to 3.80]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 0.3 [0.00 to 4.24]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.1 [0.00 to 3.81]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.1 [0.00 to 3.94]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.1 [0.00 to 3.82]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.3 [0.00 to 4.29]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.2 [0.00 to 4.09]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

34. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleeding Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time, All Emicizumab Participants
Description: as for outcome 33
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: Treated spontaneous bleeds per year
Arm/Group | All Emicizumab Participants
Number analyzed (Participants) | 151
Treated spontaneous bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 150
  1 to 12 Weeks | 0.0 [0.00 to 0.00]
  13 to 24 Weeks: number analyzed (Participants) | 148
  13 to 24 Weeks | 0.0 [0.00 to 0.00]
  25 to 36 Weeks: number analyzed (Participants) | 144
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 144
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 142
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 140
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 140
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 131
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 117
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 104
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 99
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 94
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 93
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 89
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 85
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 83
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 82
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 80
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 76
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 72
  229 to 240 Weeks | 0.0 [0.00 to 0.00]
  241 to 252 Weeks: number analyzed (Participants) | 67
  241 to 252 Weeks | 0.0 [0.00 to 0.00]
  253 to 264 Weeks: number analyzed (Participants) | 58
  253 to 264 Weeks | 0.0 [0.00 to 0.00]
  265 to 276 Weeks: number analyzed (Participants) | 22
  265 to 276 Weeks | 0.0 [0.00 to 0.00]
  277 to 288 Weeks: number analyzed (Participants) | 5
  277 to 288 Weeks | 0.0 [0.00 to 0.00]

35. Secondary Outcome: Percentage of Participants With Anti-Emicizumab Antibodies at Any Time Post-Baseline During the Study
Description: A validated enzyme-linked immunosorbent assay (ELISA) method was used to analyze the levels of anti-drug antibodies (ADAs) against emicizumab in plasma. A sample was considered positive for anti-emicizumab antibodies if the test result reached or exceeded a pre-determined threshold. 'Total ADA Positive' is the sum of all subjects who tested positive for ADA in the 2 following categories: 'ADA Positive (Treatment Boosted)', those who are pre-dose ADA positive and have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement; and 'ADA Positive (Treatment Induced)', those who are pre-dose ADA negative or missing data and who have at least one post-dose ADA positive sample.
Time Frame: From Baseline to discontinuation from study (median [min-max] observation period for all emicizumab participants: 262.3 [14.4-288.3] weeks)
Population: The All Emicizumab Population includes all participants in Arms A, B, C (Emi), and D treated with emicizumab; 1 was excluded from Arm C (Emi) (lost to follow-up before Week 24 and had not switched to emicizumab).
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
percentage of participants
  Total ADA Positive (Boosted+Induced) | 8.3 | 5.7 | 0.0 | 1.6 | 4.0
  ADA Positive (Treatment Boosted) | 0.0 | 2.9 | 0.0 | 0.0 | 0.7
  ADA Positive (Treatment Induced) | 8.3 | 2.9 | 0.0 | 1.6 | 3.3

36. Secondary Outcome: Percentage of Participants With De Novo Development of Factor VIII (FVIII) Inhibitors
Description: Levels of anti-FVIII antibodies (inhibitors) were analyzed using a validated FVIII activity assay. A participant was considered to have developed de novo FVIII inhibitors if the inhibitor levels detected in a post-baseline sample reached or exceeded a pre-determined threshold.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | All Emicizumab Participants
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 151
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

37. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Emicizumab
Description: Trough plasma concentrations of emicizumab were analyzed using a validated Enzyme Linked Immunosorbent Assay (ELISA). The lower limit of quantification (LLOQ) was 100 nanograms per milliliter (ng/mL). Because participants in Arm C (Control) switched from no prophylaxis to start receiving emicizumab prophylaxis after Week 24, the timepoints for Arm C (Emi) are expressed relative to first emicizumab dose.
Time Frame: Predose at Weeks 1, 2, 3, 4, 5, 7, 9, 13, 17, 21, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, 169, 181, 193, 205, 217, 229, 241, 253, 265, and 277
Population: The Pharmacokinetics (PK) Population includes all participants in Arms A, B, C (Emi), and D treated with emicizumab who had at least one post-dose emicizumab concentration result; 1 was excluded from Arm C (Emi) (lost to follow-up before Week 24 and had not switched to emicizumab). Number analyzed represents participants per study arm with available samples at each specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Groups:
- Arms A and D: Emicizumab 1.5 mg/kg QW: This analysis set is a combination of all emicizumab-treated participants from Arms A and D who received the same emicizumab prophylaxis dosing regimen at a dose of 3 milligrams per kilogram (mg/kg) subcutaneously (SC) once per week (QW) for 4 weeks, followed by 1.5 mg/kg emicizumab SC QW until discontinuation from the study.
- Arms B and C (Emi): Emicizumab 3 mg/kg Q2W: This analysis set is a combination of all emicizumab-treated participants from Arms B and C (Emi) who received the same emicizumab prophylaxis dosing regimen at a dose of 3 milligrams per kilogram (mg/kg) subcutaneously (SC) once per week (QW) for 4 weeks, followed by 3 mg/kg emicizumab SC once every 2 weeks (Q2W) until discontinuation from the study.
Arm/Group | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) | Arms A and D: Emicizumab 1.5 mg/kg QW | Arms B and C (Emi): Emicizumab 3 mg/kg Q2W
Number analyzed (Participants) | 36 | 35 | 17 | 63 | 99 | 52
micrograms per milliliter (μg/mL)
  Week 1: number analyzed (Participants) | 35 | 35 | 17 | 61 | 96 | 52
  Week 1 | NA (NA) — No results available because the samples were below the limit of quantification (BLQ). | NA (NA) — No results available because the samples were below the limit of quantification (BLQ). | NA (NA) — No results available because the samples were below the limit of quantification (BLQ). | NA (NA) — No results available because the samples were below the limit of quantification (BLQ). | NA (NA) — No results available because the samples were below the limit of quantification (BLQ). | NA (NA) — No results available because the samples were below the limit of quantification (BLQ).
  Week 2: number analyzed (Participants) | 36 | 35 | 17 | 62 | 98 | 52
  Week 2 | 16.3 (6.1) | 16.8 (5.9) | 19.6 (8.2) | 17.3 (5.4) | 16.9 (5.7) | 17.7 (6.8)
  Week 3: number analyzed (Participants) | 36 | 35 | 17 | 62 | 98 | 52
  Week 3 | 29.1 (9.3) | 29.2 (6.5) | 33.0 (12.6) | 30.5 (8.7) | 30.0 (8.9) | 30.5 (9.0)
  Week 4: number analyzed (Participants) | 36 | 35 | 17 | 62 | 98 | 52
  Week 4 | 41.9 (11.8) | 41.4 (9.7) | 47.9 (15.0) | 42.4 (9.4) | 42.2 (10.3) | 43.6 (11.9)
  Week 5: number analyzed (Participants) | 34 | 35 | 17 | 62 | 96 | 52
  Week 5 | 48.0 (13.7) | 48.8 (12.3) | 59.6 (20.7) | 54.5 (12.5) | 52.2 (13.2) | 52.4 (16.2)
  Week 7: number analyzed (Participants) | 32 | 33 | 17 | 61 | 93 | 50
  Week 7 | 47.9 (16.1) | 48.4 (11.4) | 55.2 (16.2) | 52.4 (13.3) | 50.9 (14.4) | 50.7 (13.5)
  Week 9: number analyzed (Participants) | 33 | 34 | 17 | 63 | 96 | 51
  Week 9 | 49.0 (16.4) | 46.4 (14.1) | 53.1 (15.7) | 55.1 (16.1) | 53.0 (16.4) | 48.7 (14.9)
  Week 13: number analyzed (Participants) | 33 | 34 | 17 | 63 | 96 | 51
  Week 13 | 48.7 (18.3) | 47.6 (16.0) | 47.9 (18.1) | 55.0 (15.9) | 52.8 (16.9) | 47.7 (16.5)
  Week 17: number analyzed (Participants) | 33 | 34 | 17 | 62 | 95 | 51
  Week 17 | 54.3 (24.0) | 48.9 (17.7) | 43.4 (16.2) | 55.0 (16.5) | 54.7 (19.3) | 47.0 (17.2)
  Week 21: number analyzed (Participants) | 32 | 34 | 16 | 61 | 93 | 50
  Week 21 | 50.7 (20.2) | 47.3 (15.5) | 45.6 (18.8) | 55.1 (16.2) | 53.6 (17.7) | 46.7 (16.4)
  Week 25: number analyzed (Participants) | 31 | 34 | 17 | 58 | 89 | 51
  Week 25 | 50.5 (21.7) | 47.6 (18.9) | 51.8 (23.4) | 54.8 (16.8) | 53.3 (18.7) | 49.0 (20.4)
  Week 33: number analyzed (Participants) | 30 | 34 | 16 | 58 | 88 | 50
  Week 33 | 56.3 (25.3) | 52.9 (22.4) | 52.0 (21.3) | 59.1 (18.5) | 58.1 (20.9) | 52.6 (21.9)
  Week 41: number analyzed (Participants) | 31 | 34 | 17 | 58 | 89 | 51
  Week 41 | 54.8 (24.2) | 48.4 (18.8) | 50.7 (24.4) | 59.6 (21.4) | 57.9 (22.4) | 49.2 (20.6)
  Week 49: number analyzed (Participants) | 31 | 32 | 17 | 58 | 89 | 49
  Week 49 | 55.4 (22.9) | 52.2 (20.2) | 54.3 (21.3) | 60.2 (19.9) | 58.5 (21.0) | 52.9 (20.4)
  Week 61: number analyzed (Participants) | 31 | 33 | 17 | 57 | 88 | 50
  Week 61 | 55.3 (21.4) | 52.0 (21.1) | 52.5 (19.8) | 61.1 (22.5) | 59.1 (22.1) | 52.2 (20.5)
  Week 73: number analyzed (Participants) | 31 | 32 | 15 | 57 | 88 | 47
  Week 73 | 54.4 (21.5) | 51.6 (21.3) | 47.8 (18.4) | 58.5 (19.2) | 57.1 (20.0) | 50.4 (20.3)
  Week 85: number analyzed (Participants) | 31 | 32 | 13 | 55 | 86 | 45
  Week 85 | 48.8 (17.4) | 46.4 (20.4) | 47.7 (17.9) | 56.7 (18.5) | 53.8 (18.5) | 46.8 (19.5)
  Week 97: number analyzed (Participants) | 28 | 29 | 11 | 48 | 76 | 40
  Week 97 | 52.6 (20.0) | 50.9 (21.0) | 51.7 (28.3) | 58.5 (18.7) | 56.3 (19.3) | 51.1 (22.9)
  Week 109: number analyzed (Participants) | 26 | 26 | 11 | 39 | 65 | 37
  Week 109 | 53.9 (19.2) | 52.3 (19.5) | 46.4 (27.0) | 59.0 (19.1) | 57.0 (19.1) | 50.5 (21.7)
  Week 121: number analyzed (Participants) | 23 | 24 | 10 | 37 | 60 | 34
  Week 121 | 58.8 (21.1) | 55.0 (22.0) | 50.0 (25.2) | 57.1 (18.2) | 57.7 (19.2) | 53.5 (22.7)
  Week 133: number analyzed (Participants) | 23 | 23 | 10 | 34 | 57 | 33
  Week 133 | 55.3 (26.0) | 54.7 (18.5) | 54.6 (26.9) | 59.3 (19.2) | 57.7 (22.1) | 54.7 (20.9)
  Week 145: number analyzed (Participants) | 23 | 22 | 6 | 33 | 56 | 28
  Week 145 | 54.1 (23.7) | 51.3 (17.7) | 44.8 (11.6) | 55.7 (20.4) | 55.0 (21.6) | 49.9 (16.6)
  Week 157: number analyzed (Participants) | 19 | 21 | 9 | 30 | 49 | 30
  Week 157 | 57.6 (27.8) | 52.2 (21.4) | 46.8 (24.0) | 55.9 (23.7) | 56.6 (25.1) | 50.6 (21.9)
  Week 169: number analyzed (Participants) | 16 | 16 | 8 | 22 | 38 | 24
  Week 169 | 53.9 (21.8) | 50.3 (19.6) | 45.8 (20.6) | 56.4 (18.0) | 55.3 (19.4) | 48.8 (19.6)
  Week 181: number analyzed (Participants) | 15 | 11 | 8 | 17 | 32 | 19
  Week 181 | 59.8 (24.8) | 48.8 (22.1) | 43.5 (26.2) | 57.5 (21.3) | 58.6 (22.7) | 46.5 (23.4)
  Week 193: number analyzed (Participants) | 17 | 18 | 7 | 21 | 38 | 25
  Week 193 | 53.9 (21.0) | 52.4 (24.6) | 42.1 (19.1) | 60.5 (19.6) | 57.5 (20.2) | 49.5 (23.3)
  Week 205: number analyzed (Participants) | 18 | 20 | 8 | 23 | 41 | 28
  Week 205 | 53.5 (20.8) | 51.9 (22.4) | 54.2 (31.1) | 58.6 (24.1) | 56.4 (22.6) | 52.6 (24.6)
  Week 217: number analyzed (Participants) | 16 | 19 | 9 | 26 | 42 | 28
  Week 217 | 54.4 (20.8) | 55.0 (20.6) | 50.8 (26.1) | 60.8 (23.2) | 58.3 (22.2) | 53.6 (22.1)
  Week 229: number analyzed (Participants) | 17 | 17 | 9 | 26 | 43 | 26
  Week 229 | 54.9 (20.9) | 47.9 (18.9) | 53.5 (30.4) | 54.4 (19.3) | 54.6 (19.7) | 49.8 (23.1)
  Week 241: number analyzed (Participants) | 16 | 18 | 6 | 24 | 40 | 24
  Week 241 | 51.9 (19.3) | 50.2 (16.8) | 52.0 (36.1) | 60.1 (23.3) | 56.8 (21.9) | 50.6 (22.2)
  Week 253: number analyzed (Participants) | 15 | 15 | 4 | 22 | 37 | 19
  Week 253 | 58.6 (28.7) | 46.5 (17.8) | 40.3 (43.9) | 58.4 (24.7) | 58.5 (26.0) | 45.2 (23.9)
  Week 265: number analyzed (Participants) | 10 | 13 | 0 | 17 | 27 | 13
  Week 265 | 58.7 (25.8) | 47.3 (14.5) |  | 60.0 (23.9) | 59.5 (24.2) | 47.3 (14.5)
  Week 277: number analyzed (Participants) | 6 | 5 | 0 | 2 | 8 | 5
  Week 277 | 71.9 (34.2) | 49.0 (16.2) |  | 61.3 (17.2) | 69.2 (30.1) | 49.0 (16.2)

ADVERSE EVENTS:
Time Frame: Total observation time for all participants: From enrollment until study completion (median [min-max] 262.3 [14.4-288.3] weeks); Arm C (Control): From enrollment to 24 weeks on no prophylaxis (median [min-max]: 24.00 [14.4-25.0] weeks)
Description: All adverse events (AEs) in emicizumab-treated subjects are reported, including after dose up-titration or change of dosing regimen. AEs in Arm C are reported in 2 groups: Arm C (Control) for the first 24 weeks on no prophylaxis; Arm C (Emi) for those who switched after 24 weeks to receive emicizumab prophylaxis.
Groups:
- Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis): This arm includes all participants from Arm C who had switched to emicizumab prophylaxis during the entire study after having completed 24 weeks on No Prophylaxis. The data reported was collected only during emicizumab prophylaxis treatment. Emicizumab was administered at a loading dose of 3 mg/kg SC once per week (QW) for the first 4 weeks, followed by maintenance dosing of 3 mg/kg emicizumab SC Q2W. Upon implementation of protocol version 4 (20-Dec-2019), treatment duration was extended. During this study prolongation, each participant was given the option to choose a preferred emicizumab dosing regimen among those permitted and continue on that dosing regimen until discontinuation from the study.
Arm/Group | Arm C (Control): No Prophylaxis | Arm A: Emicizumab 1.5 mg/kg QW | Arm B: Emicizumab 3 mg/kg Q2W | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/36 | 0/35 | 0/17 | 0/63
Serious Adverse Events (participants affected / at risk) | 1/18 | 10/36 | 8/35 | 1/17 | 16/63
Other Adverse Events (participants affected / at risk) | 5/18 | 35/36 | 33/35 | 15/17 | 61/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Control): No Prophylaxis (N=18) | Arm A: Emicizumab 1.5 mg/kg QW (N=36) | Arm B: Emicizumab 3 mg/kg Q2W (N=35) | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) (N=17) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) (N=63)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPLENIC ARTERY ANEURYSM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GINGIVAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBPERIOSTEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
DURAL TEAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BONE GIANT CELL TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PUTAMEN HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE LOOSENING (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RENAL HAEMATOMA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Control): No Prophylaxis (N=18) | Arm A: Emicizumab 1.5 mg/kg QW (N=36) | Arm B: Emicizumab 3 mg/kg Q2W (N=35) | Arm C (Emi): Emicizumab 3 mg/kg Q2W (Switch From No Prophylaxis) (N=17) | Arm D: Emicizumab 1.5 mg/kg QW (Pre-study FVIII Prophylaxis) (N=63)
HYDROCELE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 3 (4) | 2 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 4 (4) | 5 (6) | 2 (3) | 6 (6)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 7 (9)
VOMITING (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (5)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
INJECTION SITE REACTION (General disorders) | 0 (0) | 10 (37) | 8 (25) | 4 (4) | 24 (42)
PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 6 (7)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BODY TINEA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 3 (4)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
CORONAVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 7 (7)
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
GASTRIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 7 (8) | 4 (4) | 2 (2) | 9 (10)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 9 (16) | 8 (19) | 3 (4) | 20 (35)
PERIODONTITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (10)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 8 (11) | 6 (9) | 3 (4) | 14 (19)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (5)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 3 (15) | 2 (3) | 2 (3) | 6 (13)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 8 (9)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 5 (9)
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 10 (17)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 3 (5)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
TONGUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 5 (5)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 16 (41) | 11 (26) | 3 (5) | 25 (78)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (11) | 3 (4) | 2 (3) | 8 (10)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
HAEMOPHILIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (10)
MUSCLE CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 6 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 4 (4) | 0 (0) | 6 (7)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 7 (9)
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 7 (13) | 7 (30) | 2 (2) | 14 (33)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 4 (7)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 7 (9)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (12)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (5)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 9 (9)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02847637/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02847637/SAP_001.pdf